CLINICAL TRIAL: NCT02431143
Title: An Open-label Clinical Trial to Assess the Pharmacokinetics and Safety of Miltefosine Allometric Dose for the Treatment of Children With Primary Visceral Leishmaniasis in Eastern Africa
Brief Title: Pharmacokinetics/Safety of Miltefosine Allometric Dose for the Treatment of Visceral Leishmaniasis in Children in Eastern Africa
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Drugs for Neglected Diseases (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LEAP 0714
Record Dates: First submitted 2015-04-20; First posted 2015-04-30 (Estimated); Last update posted 2016-10-11 (Estimated); Status verified 2016-10

CONDITIONS: Visceral Leishmaniasis
MeSH Terms: conditions — Leishmaniasis, Visceral | interventions — miltefosine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Miltefosine (Experimental): allometric dosing
  Interventions: Drug: Miltefosine

INTERVENTIONS:
Drug: Miltefosine

SUMMARY:
This is a multicenter, non-comparative, open-label clinical trial to assess the Pharmacokinetics (PK) and safety of miltefosine using an allometric dose algorithm in the treatment of children with primary Visceral Leishmaniasis (VL) in eastern Africa. Efficacy and Pharmacodynamics (PD) will be assessed as secondary outcomes.

The proposed study aims to assess whether drug exposure in children can be increased to equivalent adult drug exposure by using the miltefosine allometric dose given BID for 28 days in paediatric VL patients aged 4-12y and whether this dose is tolerable. The present study is also expected to provide the basis for minimum time to reach sufficient drug exposure for miltefosine activity to guide optimal treatment duration to be used in combination therapy for visceral leishmaniasis. The PK data will be assessed in this trial using a compartmental population PK approach.

ELIGIBILITY:
Inclusion Criteria:

* Patients with clinical signs and symptoms of VL and confirmatory parasitological microscopic diagnosis
* Patients aged > 4 to < 12 years who are able to comply with the study protocol.
* Patients for whom written informed consent has been signed by parents(s) or legal guardian
* Weight < 30 kg

Exclusion Criteria:

* Patients who are relapse cases
* Patients who have received any anti-leishmanial drugs in the last 6 months
* Patients with severe malnutrition (for children aged <5 years, weight-for-height WHO reference curves by gender, z score <-3; for children 5-12 years, BMI-for-age WHO reference curves for gender, z score < -3)
* Patients with positive HIV diagnosis
* Patients with previous history of hypersensitivity reaction to miltefosine
* Patients suffering from a concomitant severe infection such as Tuberculosis (TB) or any other serious underlying disease (cardiac, renal, hepatic) which would preclude evaluation of the patient's response to study medication
* Patients suffering from other conditions associated with splenomegaly such as schistosomiasis
* Pregnant or lactating women or female patient in childbearing age (reached menarche)
* Patients with haemoglobin < 5g/dl
* Patients with White Blood Cells (WBC) < 1 x 10³/mm³
* Patients with platelets < 40,000/mm³
* Patients with abnormal liver function (ALT and AST) tests of more than three times the normal range.
* Patients with bilirubin more than 1.5 times the upper normal range
* Patients with serum creatinine above the upper limit of normal (ULN) for age and gender.
* Patients with clinical signs of severe VL disease such as jaundice and bleeding
* Patients who cannot comply with the planned scheduled visits and procedures of the study protocol

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2015-05; Primary Completion 2016-04 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics Parameters (Area Under the Curve (AUC) - composite outcome) | During treatment, at 1 and 6 months follow-up
  Area Under the Curve calculation is based on several timepoints from first drug intake up to complete elimination of the drug.
Safety (composite outcome) adverse events | until day 210
  1. Frequency of Serious Adverse Events (SAEs) and Adverse Events (AEs) requiring treatment discontinuation, 2. Frequency and severity of adverse events
Pharmacokinetics Parameters (Css/Cmax) | Day 28

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Rashid Juma, MD, Principal Investigator — Kenya Medical Research Institute
Locations (2):
- Kacheliba Hospital, Kacheliba, Rift Valley, West Pokot, Kenya
- Amudat Hospital, Amudat, Karamoja, Uganda

REFERENCES:
- [Derived] Mbui J, Olobo J, Omollo R, Solomos A, Kip AE, Kirigi G, Sagaki P, Kimutai R, Were L, Omollo T, Egondi TW, Wasunna M, Alvar J, Dorlo TPC, Alves F. Pharmacokinetics, Safety, and Efficacy of an Allometric Miltefosine Regimen for the Treatment of Visceral Leishmaniasis in Eastern African Children: An Open-label, Phase II Clinical Trial. Clin Infect Dis. 2019 Apr 24;68(9):1530-1538. doi: 10.1093/cid/ciy747. PMID 30188978